CLINICAL TRIAL: NCT01080521
Title: A Prospective Study of Cognitive Function During Chemotherapy for Front-Line Treatment of Ovarian, Primary Peritoneal or Fallopian Tube Cancer
Brief Title: Changes in Brain Function in Patients With Stage I, Stage II, Stage III, or Stage IV Ovarian, Primary Peritoneal, or Fallopian Tube Cancer Who Are Receiving Chemotherapy
Status: Completed | Type: Observational
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Other Study IDs: GOG-0256; NCI-2011-02213 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-0256; CDR0000666786; GOG-0256 (Other: Gynecologic Oncology Group); GOG-0256 (Other: DCP); GOG-0256 (Other: CTEP); U10CA101165 (NIH)
Record Dates: First submitted 2010-03-03; First posted 2010-03-04 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Cognitive Side Effects of Cancer Therapy; Malignant Ovarian Epithelial Tumor; Ovarian Brenner Tumor; Ovarian Carcinosarcoma; Ovarian Choriocarcinoma; Ovarian Clear Cell Cystadenocarcinoma; Ovarian Dysgerminoma; Ovarian Embryonal Carcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Mixed Germ Cell Tumor; Ovarian Mucinous Cystadenocarcinoma; Ovarian Polyembryoma; Ovarian Sarcoma; Ovarian Seromucinous Carcinoma; Ovarian Serous Cystadenocarcinoma; Ovarian Teratoma; Ovarian Yolk Sac Tumor; Stage I Ovarian Cancer; Stage IA Fallopian Tube Cancer; Stage IA Ovarian Cancer; Stage IA Ovarian Germ Cell Tumor; Stage IB Fallopian Tube Cancer; Stage IB Ovarian Cancer; Stage IB Ovarian Germ Cell Tumor; Stage IC Fallopian Tube Cancer; Stage IC Ovarian Cancer; Stage IC Ovarian Germ Cell Tumor; Stage II Ovarian Cancer; Stage IIA Fallopian Tube Cancer; Stage IIA Ovarian Cancer; Stage IIA Ovarian Germ Cell Tumor; Stage IIB Fallopian Tube Cancer; Stage IIB Ovarian Cancer; Stage IIB Ovarian Germ Cell Tumor; Stage IIC Fallopian Tube Cancer; Stage IIC Ovarian Cancer; Stage IIC Ovarian Germ Cell Tumor; Stage IIIA Fallopian Tube Cancer; Stage IIIA Ovarian Cancer; Stage IIIA Ovarian Germ Cell Tumor; Stage IIIA Primary Peritoneal Cancer; Stage IIIB Fallopian Tube Cancer; Stage IIIB Ovarian Cancer; Stage IIIB Ovarian Germ Cell Tumor; Stage IIIB Primary Peritoneal Cancer; Stage IIIC Fallopian Tube Cancer; Stage IIIC Ovarian Cancer; Stage IIIC Ovarian Germ Cell Tumor; Stage IIIC Primary Peritoneal Cancer; Stage IV Fallopian Tube Cancer; Stage IV Ovarian Cancer; Stage IV Ovarian Germ Cell Tumor; Stage IV Primary Peritoneal Cancer; Undifferentiated Ovarian Carcinoma
MeSH Terms: conditions — Brenner Tumor; Dysgerminoma; Teratoma, Ovarian; Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Observational (cognitive function during chemotherapy): Patients receive standard chemotherapy. Treatment repeats for 6 courses. Patients complete neurocognitive evaluations (Patient Assessment and Own Functioning scale and HeadMinder Custom Research Tool) and quality-of-life assessments (Hospital Anxiety and Depression Scale, FACT-O, and FACT/GOG-Ntx subscale) at baseline, before the fourth course of chemotherapy, at 3 weeks after the sixth course of chemotherapy, and at 6 months after the sixth course of chemotherapy.
  Interventions: Procedure: Cognitive Assessment; Other: Quality-of-Life Assessment

INTERVENTIONS:
Procedure: Cognitive Assessment — Ancillary studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This clinical trial is studying changes in brain function in patients with stage I, stage II, stage III, or stage IV ovarian, primary peritoneal, or fallopian tube cancer who are receiving chemotherapy. Learning about the effects of chemotherapy on brain function may help doctors plan cancer treatments.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To describe changes in cognitive function among patients with ovarian, primary peritoneal, or fallopian tube cancer receiving front-line chemotherapy as measured by a web-based assessment of cognitive function as measured by the HeadMinder Customized Research Tool (CRT).

SECONDARY OBJECTIVES:

I. To estimate the proportion of these patients who experience possible or probable acute or persistent impairment in cognitive function while receiving chemotherapy as measured by a web-based assessment of cognitive function as measured by the HeadMinder CRT.

II. To explore the association between the patient-reported neurocognitive function as measured by the Patient Assessment of Own Functioning (PAF) scale and web-based assessment of cognitive function as measured by the HeadMinder CRT.

TERTIARY OBJECTIVES:

I. To explore the relationship between patient-reported quality of life as measured by the FACT-O and cognitive function as measured by the web-based and patient-reported assessments, respectively. (Exploratory) II. To explore whether the patient-reported cognitive function or the web-based assessment of cognitive function is associated with anxiety and depression as measured by the Hospital Anxiety and Depression Scale. (Exploratory) III. To explore the changes in cognitive function using the web-assessed (CRT) and self-reported (PAF) assessments, respectively, among patients with advanced ovarian cancer (stage III-IV, optimally debulked disease at enrollment) receiving IV as compared to intraperitoneal treatment. (Exploratory) IV. To explore whether the cognitive impairment as measured with web-based assessment is associated with patient age, hemoglobin, platelet count, patient-reported neurotoxicity symptoms as measured with FACT/GOG-Ntx subscale, or body weight. (Exploratory)

OUTLINE: This is a multicenter study.

Patients receive standard chemotherapy. Treatment repeats for 6 courses. Patients complete neurocognitive evaluations (Patient Assessment and Own Functioning scale and HeadMinder Custom Research Tool) and quality-of-life assessments (Hospital Anxiety and Depression Scale, FACT-O, and FACT/GOG-Ntx subscale) at baseline, before the fourth course of chemotherapy, at 3 weeks after the sixth course of chemotherapy, and at 6 months after the sixth course of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or pathologically confirmed primary diagnosis of stage I-IV ovarian, primary peritoneal, or fallopian tube cancer (any cell type)
* Planning to receive ≥ 6 courses of front-line chemotherapy

  * Have not yet received the first course of chemotherapy
* GOG performance status 0-2
* Able to read and understand English
* No uncontrolled or severe cardiovascular disease, including any of the following:

  * Myocardial infarction within the past year
  * Uncontrolled hypertension
  * Congestive heart failure
* No history of head injury with GCS < 13
* No severe hemiparesis or other condition preventing bimanual keyboard operation
* No distal neuropathy, action tremor, or other motor dysfunction that would substantially decrease keyboard accuracy
* No severe motor or mental slowing (i.e., patient who is disoriented/level C on any criterion as assessed by the person-place-time criteria)
* No other invasive malignancies within the past 5 years except for nonmelanoma skin cancer
* More than 6 months since prior epoetin alfa, darbepoetin, or any investigational forms of erythropoietin

  * Patients may receive these agents during chemotherapy treatment as needed
* No prior radiotherapy or chemotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients With Stage I, Stage II, Stage III, or Stage IV Ovarian, Primary Peritoneal, or Fallopian Tube Cancer Who Are Receiving Chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 247 (Actual)
Dates: Start 2010-04; Primary Completion 2012-01 (Actual); Study Completion 2018-01-27 (Actual)

PRIMARY OUTCOMES:
Cognitive function as measured by the HeadMinder Customized Research Tool (CRT) | Up to 6 months after completion of chemotherapy

SECONDARY OUTCOMES:
Patient-reported cognitive function as measured by Patient Assessment Own Functioning scale and web CRT | Up to 6 months after completion of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Hess, Principal Investigator — Gynecologic Oncology Group
Locations (182):
- United States (182):
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Roy and Patricia Disney Family Cancer Center, Burbank, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - University of California San Diego, San Diego, California
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Florida Hospital Orlando, Orlando, Florida
  - John B Amos Cancer Center, Columbus, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Northwestern University, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Shawnee Mission Medical Center-KCCC, Shawnee Mission, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - Baystate Medical Center, Springfield, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Michiana Hematology Oncology PC-Niles, Niles, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - Saint Dominic-Jackson Memorial Hospital, Jackson, Mississippi
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hosiptal, Pinehurst, North Carolina
  - Duke Raleigh Hospital, Raleigh, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Akron General Medical Center, Akron, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Gynecologic Oncology Group, Philadelphia, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Cancer Centers of the Carolinas-Greer Medical Oncology, Greer, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Parkland Memorial Hospital, Dallas, Texas
  - Clements University Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Virginia Mason CCOP, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Marshfield Clinic at James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Clinic Cancer Care at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin